CLINICAL TRIAL: NCT06250582
Title: Does Virtual Reality Improve Symptom Burden in Dialysis Patients?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Blum (Other)
Responsible Party: Sponsor-Investigator, David Blum, Head of the department for Palliative Care of the University hospital Zurich, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00900
Record Dates: First submitted 2023-12-20; First posted 2024-02-09 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Dialysis; Virtual Reality
MeSH Terms: interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality therapy, then standard of care (Experimental): During the intervention phase (A) participants will receive virtual reality therapy during their dialysis sessions over a period of one month. After a washout phase of one week, participants will run through a control phase (B, standard of care) also for a period of one month. Subjects will be randomized to an AB or BA sequence.
  Interventions: Other: virtual reality therapy
- standard of care, then virtual reality therapy (Experimental): During the control phase (B) participants will be treated according to standard of care over a period of one mont. After a washout phase of one week, participants will run through an intervention phase (A) and will receive virtual reality therapy during their dialysis sessions. Also for a period of one month. Subjects will be randomized to an AB or BA sequence.
  Interventions: Other: virtual reality therapy

INTERVENTIONS:
Other: virtual reality therapy — A virtual reality therapy will be applied for 30 minutes. Patients will be wearing the glasses while lying in bed/chair during their regular dialysis session. Vital signs will be monitored repeatedly. At defined times, patients are asked to answer various questionnaires about their physical and mental health.

SUMMARY:
The goal of this clinical trial is to investigate the use of virtual reality therapy in dialysis patients. The main question it aims to answer is: Does virtual reality improve symptom burden in dialysis patients and improve their mental wellbeing? Over a period of one month, one virtual reality therapy session of 30 minutes will be performed during each regular hemodialysis session. Since we will conduct a monocentric, crossover randomized controlled trial, the participants act as their own control group.

DETAILED DESCRIPTION:
Hemodialysis is a lifesaving therapy for patients with end stage kidney disease but comes with a high burden of physical and emotional symptoms that lower quality of life in dialysis patients. Dialysis mediated complications such as drops in blood pressure, nausea and muscle cramps results in refusal and a negative perception of this treatment. In dialysis patients, treatment-related burden results in deterioration in health related quality of life. During the past few years, Virtual reality (VR) has become more affordable and found its way into households as entertainment electronics but stepwise also into medicine. VR enables the user to view, interact and be immersed in a multisensory 3D virtual world. The aim of the current study is to reduce dialysis-related burden of symptoms by using virtual reality therapy during regular dialysis sessions and thereby improve quality of life among dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years;
* in treatment with thrice-weekly hemodialysis sessions;
* regular hemodialysis duration of three to five hours
* having no visual impairment
* having no acoustic deficit
* patient must be capable of speaking and understanding German or English
* no signs of cognitive impairment
* patient oriented in time and space
* being able to give informed consent as documented by signature

Exclusion Criteria:

* diagnosis of epilepsy
* current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of symptom burden of dialysis patients and improvement of their mental wellbeing | 10 weeks
  questionnaire

SECONDARY OUTCOMES:
Evaluation of the effects of virtual reality therapy during hemodialysis on heart rate | 10 weeks
  Heart rate (beats per minute)
Evaluation of the effects of virtual reality therapy during hemodialysis on blood pressure | 10 weeks
  Blood pressure (mm Hg)
To assess the acceptability and appropriateness of using VRT during hemodialysis from the perspectives of patients | 10 weeks
  questionnaire
To assess the acceptability and appropriateness of using VRT during hemodialysis from the perspectives of clinical staff | 10 weeks
  questionnaire
To test the internal consistency of the ESAS-r: Renal Score | 10 weeks
  Cronbach's alpha

CONTACTS AND LOCATIONS:
Overall Officials: David Blum, Prof. Dr., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No